CLINICAL TRIAL: NCT06380179
Title: Assessing the Impact of Post-Exercise Photobiomodulation Application on Performance, Recovery, and Behavioral State in Trained Special Operator Population
Brief Title: Photomedicine Project 14: PBMT for Performance Enhancement in SOF
Acronym: SOF
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Musculoskeletal Injury Rehabilitation Research for Operational Readiness (MIRROR) (Unknown)
Collaborators: Uniformed Services University (USU) of the Health Sciences (Unknown); 1st Special Forces Group (Airborne), United States Army (Unknown); United States Army Special Operations Command (Unknown); The Geneva Foundation (Other)
Responsible Party: Sponsor
Organization: Musculoskeletal Injury Rehabilitation Research for Operational Readiness (U.S. Federal Agency)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: USUHS.2023-126
Record Dates: First submitted 2024-03-13; First posted 2024-04-23 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-07

CONDITIONS: Photobiomodulation Therapy; Photomedicine; Low-Level Laser Therapy; Performance Enhancement; Quadriceps; Special Operations Readiness
MeSH Terms: interventions — Low-Level Light Therapy

STUDY DESIGN:
Intervention Model Description: Approach: Special Operators attending THOR3 coach led training will be invited to participate. After consenting and screening for inclusion/exclusion, participants will be randomized into two groups: 1) sham PBMT and 2) PBMT (applied to quadriceps up to 3 times per week, post coach-led training, taking approximately 5-20 minutes each time). Baseline measurements will include body fat percentage, height, weight and military/demographic information. Metrics for counter movement jump and self-reported delayed muscle onset soreness will be taken at baseline and weekly for three weeks. Isokinetic dynamometer measurements for the lower extremities, and self-reported exertion and fatigue will be taken at baseline and at the 3-week follow-up (post three-week intervention). Oura rings will be assigned at baseline and will continuously measure sleep, heart rate, Sp02, and activity. Activity and pain will also be self-reported throughout the duration of the study.
Who Masked: Participant
Masking Description: In order to facilitate participant blinding to their randomized study group, all participants (regardless of their assigned study group) will be asked to wear blackout glasses and headphones during their treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Photobiomodulation Treatment (PBMT) (Active Comparator): PBMT will be delivered at 32-40 watts (W) (depending on participant skin pigmentation). PBMT will be applied to the quadriceps area. A study team member will use the quadriceps measurements of the treatment area to calculate the PBMT treatment time (approximately 5-20 minutes) and specified J/cm2. PBMT treatment will be provided 3 times per week, for 3 weeks.
  Interventions: Device: THOR3 training + Photobiomodulation Therapy (PBMT)
- Sham PBMT (Sham Comparator): The inclusion of sham PBMT will ensure all participant treatment procedures remain the same, with the exception of emission of photons (active treatment), thus, allowing for contribution of any differences between groups to be credited to the use of PBMT.
  Interventions: Device: THOR3 training + sham PBMT

INTERVENTIONS:
Device: THOR3 training + Photobiomodulation Therapy (PBMT) — PBMT will be delivered at 32-40W (depending on participant skin pigmentation). PBMT will be applied to the quadriceps area. A study team member will use the quadriceps measurements of the treatment area to calculate the PBMT treatment time (approximately 5-20 minutes) and specified J/cm2. PBMT treatment will be provided 3 times per week, for 3 weeks.
  PBMT will be delivered by a trained study team member using the LightForce® XLi 40W device with the Smart Hand Piece technology, which has a built-in accelerometer in the hand piece that controls the speed of light delivery to the treatment area. The trained team members will use the Smart Hand Piece technology, which assesses the operator's speed and provides real-time visual and sensory feedback calibrated to shut-off when moving too slowly and warns the operator when moving too quickly by vibrating. Treatment is delivered through a flexible optical fiber threaded through the hand piece, which contains a rolling glass massage ball.
  Other Names: Low-level Laser Therapy (LLLT); LightForce® XLi
  Arms: Photobiomodulation Treatment (PBMT)
Device: THOR3 training + sham PBMT — Sham PBMT will be provided by a trained study team member. Sham PBMT will be delivered in the same manner as indicated for the PBMT process above, but the device will stay in standby mode (i.e., the treatment mode will not be turned on). As infrared light is invisible to the naked eye, the only visible difference between treatment and standby modes is the presence of a few tiny amber lights (these lights are on during treatment mode).
  Other Names: THOR3 training + placebo
  Arms: Sham PBMT

SUMMARY:
Special Operations Forces (SOF) train continually to maintain peak performance. Thus, they are nearly always in a state of recovery, and in need of noninvasive therapies to address the taxing workload. Photobiomodulation therapy (PBMT) is a noninvasive treatment where a low-level laser is applied to the body to enhance healing, recovery, and performance. Army Tactical Human Optimization Rapid Rehabilitation and Reconditioning (THOR3) provides a consistent avenue for implementation of PBMT as a modality. Studies in athletes have shown performance and recovery benefits with pre-and post-workout focal application of PBMT. While there is less evidence on the potential cognitive/behavioral effects of a systematic application of PBMT, self-reported fatigue has also been found to be significantly lower in groups with focal PBMT application as compared to placebo. Further, PBMT research in healthy military tactical athletes is limited. PBMT may be a promising tool for enhancing physical performance by accelerating musculoskeletal and psychological recovery in the SOF population. The investigators aim to study the physiologic and behavioral effects of PBMT application post-exercise on performance in SOF Operators.

The Intent: The investigators propose to conduct a single-blinded randomized-control trial with sham control to investigate the effectiveness of providing PBMT post physical training in a SOF population.

The specific aims of this study are to:

1. Analyze and describe the physiologic effects, if any, of PBMT application post-exercise in Special Forces Operators undergoing coach-led training.
2. Analyze and describe the behavioral effects, if any, of PBMT application post-exercise in Special Forces Operators undergoing coach-led training.
3. Evaluate the overall clinical utility of focal PBMT subsequent to physical training in a US Army SOF, tactical athlete population.

ELIGIBILITY:
Inclusion Criteria:

* Active-Duty Special Forces Personnel (18-series)
* Able to read and understand English language for consent purposes
* Able to commit to study intervention and follow-up
* Able to participate in THOR3 coach-lead training, without restriction

Exclusion Criteria:

* Obese (body fat > 25%)
* Cardiovascular disease
* Use of select medications (e.g., statins, diuretics, hypertensive agents)
* Female
* Tattoo in treatment area (body region)
* Diagnosis with porphyria (light induced allergy) or photosensitive eczema
* Current use of medications associated with sensitivity to heat or light (e.g., amiodarone, chlorpromazine, doxycycline, hydrochlorothiazide, nalidixic acid, naproxen, piroxicam, tetracycline, thioridazine, voriconazole)
* Use of pacemaker/underlying cardiac disease
* Diagnosed with autoimmune disease(s)
* Albinism
* Peripheral Neuropathy

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Estimated)
Dates: Start 2025-01-23 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Countermovement Jump (CMJ) initial baseline: deceleration/concentric impulse | Collected prior to treatment starting at time of enrollment.
  Assesses dynamic strength performance, including deceleration/concentric impulse via force plates and analysis software.
Countermovement Jump (CMJ) initial baseline: peak force production | Collected prior to treatment starting at time of enrollment.
  Assesses dynamic strength performance, including peak force production via force plates and analysis software.
Countermovement Jump (CMJ) initial baseline: rate of force production | Collected prior to treatment starting at time of enrollment.
  Assesses dynamic strength performance, including rate of force production via force plates and analysis software.
Countermovement Jump (CMJ) initial baseline: unilateral performance comparison | Collected prior to treatment starting at time of enrollment.
  Assesses dynamic strength performance, including comparisons between unilateral lower extremity performance via force plates and analysis software.
Countermovement Jump (CMJ) week 1 follow-up: deceleration/concentric impulse | Collected at the end of week 1 prior to coach-led training.
  Assesses dynamic strength performance, including deceleration/concentric impulse via force plates and analysis software.
Countermovement Jump (CMJ) week 1 follow-up: peak force production | Collected at the end of week 1 prior to coach-led training.
  Assesses dynamic strength performance, including peak force production via force plates and analysis software.
Countermovement Jump (CMJ) week 1 follow-up: rate of force production | Collected at the end of week 1 prior to coach-led training.
  Assesses dynamic strength performance, including rate of force production via force plates and analysis software.
Countermovement Jump (CMJ) week 1 follow-up: unilateral performance comparison | Collected at the end of week 1 prior to coach-led training.
  Assesses dynamic strength performance, including comparisons between unilateral lower extremity performance via force plates and analysis software.
Countermovement Jump (CMJ) week 2 follow-up: deceleration/concentric impulse | Collected at the end of week 2 prior to coach-led training.
  Assesses dynamic strength performance, including deceleration/concentric impulse via force plates and analysis software.
Countermovement Jump (CMJ) week 2 follow-up: peak force production | Collected at the end of week 2 prior to coach-led training.
  Assesses dynamic strength performance, including peak force production via force plates and analysis software.
Countermovement Jump (CMJ) week 2 follow-up: rate of force production | Collected at the end of week 2 prior to coach-led training.
  Assesses dynamic strength performance, including rate of force production via force plates and analysis software.
Countermovement Jump (CMJ) week 2 follow-up: unilateral performance comparison | Collected at the end of week 2 prior to coach-led training.
  Assesses dynamic strength performance, including comparisons between unilateral lower extremity performance via force plates and analysis software.
Countermovement Jump (CMJ) week 3 follow-up: deceleration/concentric impulse | Collected at the end of week 3 prior to coach-led training.
  Assesses dynamic strength performance, including deceleration/concentric impulse via force plates and analysis software.
Countermovement Jump (CMJ) week 3 follow-up: peak force production | Collected at the end of week 3 prior to coach-led training.
  Assesses dynamic strength performance, including peak force production via force plates and analysis software.
Countermovement Jump (CMJ) week 3 follow-up: rate of force production | Collected at the end of week 3 prior to coach-led training.
  Assesses dynamic strength performance, including rate of force production via force plates and analysis software.
Countermovement Jump (CMJ) week 3 follow-up: unilateral performance comparison | Collected at the end of week 3 prior to coach-led training.
  Assesses dynamic strength performance, including comparisons between unilateral lower extremity performance via force plates and analysis software.
Isometric Quadriceps Strength Testing initial baseline | Collected prior to treatment starting at time of enrollment.
  Measuring isolated strength.
Isometric Hamstrings Strength Testing initial baseline | Collected prior to treatment starting at time of enrollment.
  Measuring isolated strength.
Isokinetic Quadriceps Strength Testing initial baseline | Collected prior to treatment starting at time of enrollment.
  Measuring isolated strength.
Isokinetic Hamstrings Strength Testing initial baseline | Collected prior to treatment starting at time of enrollment.
  Measuring isolated strength.
Isometric Quadriceps Strength Testing 3-week follow-up | Collected at the 3-week follow-up session prior to coach-led training.
  Measuring isolated strength.
Isometric Hamstrings Strength Testing 3-week follow-up | Collected at the 3-week follow-up session prior to coach-led training.
  Measuring isolated strength.
Isokinetic Quadriceps Strength Testing 3-week follow-up | Collected at the 3-week follow-up session prior to coach-led training.
  Measuring isolated strength.
Isokinetic Hamstrings Strength Testing 3-week follow-up | Collected at the 3-week follow-up session prior to coach-led training.
  Measuring isolated strength.
Defense and Veteran's Pain Rating Scale (DVPRS) initial baseline | Self-reported, daily from date of randomization through study completion after 3 weeks.
  Captures subjective pain rating on a 0 - 10 scale (minimum - maximum; 0 = no pain, 10 = severe pain)
Defense and Veteran's Pain Rating Scale (DVPRS) daily reports | Self-reported, daily from date of randomization through study completion after 3 weeks.
  Captures subjective pain rating on a 0 - 10 scale (minimum - maximum; 0 = no pain, 10 = severe pain)
Visual Analog Scale (VAS) initial baseline | Collected prior to treatment starting at time of enrollment.
  Measures delayed onset muscle soreness. Respondents mark on a 10 centimeter line their current level of muscle soreness. The left end of the line represents "I feel no soreness in my muscles" and the right end represents "My muscles feel so sore, I don't want to move them."
Visual Analog Scale (VAS) week 1 follow-up | Collected at the end of week 1 after coach-led training and laser treatment.
  Measures delayed onset muscle soreness. Respondents mark on a 10 centimeter line their current level of muscle soreness. The left end of the line represents "I feel no soreness in my muscles" and the right end represents "My muscles feel so sore, I don't want to move them."
Visual Analog Scale (VAS) week 2 follow-up | Collected at the end of week 2 after coach-led training and laser treatment.
  Measures delayed onset muscle soreness. Respondents mark on a 10 centimeter line their current level of muscle soreness. The left end of the line represents "I feel no soreness in my muscles" and the right end represents "My muscles feel so sore, I don't want to move them."
Visual Analog Scale (VAS) week 3 follow-up | Collected at the end of week 3 after coach-led training and laser treatment.
  Measures delayed onset muscle soreness. Respondents mark on a 10 centimeter line their current level of muscle soreness. The left end of the line represents "I feel no soreness in my muscles" and the right end represents "My muscles feel so sore, I don't want to move them."
Borg Modified Rating of Perceived Exertion (RPE) initial baseline | Collected prior to treatment starting at time of enrollment
  Quantifying perceived exertion on 0-10 scale.
Borg Modified Rating of Perceived Exertion (RPE) 3-week follow-up | Collected at the 3-week follow-up session after coach-led training and laser treatment.
  Quantifying perceived exertion on 0-10 scale.
Elloumi fatigue scale initial baseline | Collected prior to treatment starting at time of enrollment.
  Behavioral health rating of fatigue. The short questionnaire of fatigue uses eight questions that highlight perception of training difficulty, sleep, leg discomfort, infection/colds, concentration, work efficacy, anxiety and overall stress. Each question is rated by the respondent on a 7-point scale: 1 point (not at all) to 7 points (very much). The summed total score of the 8 questions allows for a total score of fatigue (TSF). Total score of fatigue ranges from 8 points (not at all fatigued) to 56 points (very much fatigued).
Elloumi fatigue scale 3-week follow-up | Collected at the 3-week follow-up session after coach-led training and laser treatment.
  Behavioral health rating of fatigue. The short questionnaire of fatigue uses eight questions that highlight perception of training difficulty, sleep, leg discomfort, infection/colds, concentration, work efficacy, anxiety and overall stress. Each question is rated by the respondent on a 7-point scale: 1 point (not at all) to 7 points (very much). The summed total score of the 8 questions allows for a total score of fatigue (TSF). Total score of fatigue ranges from 8 points (not at all fatigued) to 56 points (very much fatigued).
Quick Physical Activity Rating scale (QPAR) | Collected prior to treatment starting at time of enrollment.
  Scaled rating of various types of physical activity participation. Respondent reporting quantifies the overall amount of physical activity that the respondent regularly engages in. Activities are weighted in intensity that ranges from 1 (light) to 3 (heavy). Activity weekly frequency reported as never (0 days), seldom (1-2 days), sometime (3-4 days), and often (5-7 days). Activity duration collected as less than one hour per day, 1-2 hours per day, and more than two hours per day. Intensity (1-3), frequency (0-3) and duration (1-3) scores are multiplied and provide a physical activity score that may range from 0 - 153 points, 0 being very low physical activity and 153 representing very high physical activity.
Oura Ring Sleep Data: sleep metrics - sleep duration | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of sleep, including duration of sleep.
Oura Ring Sleep Data: sleep metrics - time in bed | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of sleep, including time spent in bed.
Oura Ring Sleep Data: sleep metrics - light sleep length | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of sleep, including duration of light sleep stage.
Oura Ring Sleep Data: sleep metrics - rapid eye movement (REM) sleep length | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of sleep, including duration of REM sleep stage.
Oura Ring Sleep Data: sleep metrics - deep sleep length | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of sleep, including duration of deep sleep stage.
Oura Ring Sleep Data: sleep metrics - sleep latency | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of sleep, including sleep latency (time taken to fall asleep).
Oura Ring Sleep Data: sleep metrics - sleep efficiency score | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of sleep, including sleep efficiency score.
Oura Ring Sleep Data: sleep metrics - sleep quality score | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of sleep, including sleep quality score.
Oura Ring Sleep Data: Readiness trends - body temperature changes | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of physical readiness trends, including changes in body temperature.
Oura Ring Sleep Data: Readiness trends - heart rate changes | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of physical readiness trends, including changes in heart rate.
Oura Ring Sleep Data: Readiness trends - heart rate variability (HRV) | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of physical readiness trends, including HRV - a measure of the fluctuation in the time intervals between adjacent heartbeats.
Oura Ring Sleep Data: Readiness trends - respiration rate | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of physical readiness trends, including respiratory rate.
Oura Ring Sleep Data: Readiness trends - blood oxygen saturation | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of physical readiness trends, including blood oxygen saturation.
Oura Ring Sleep Data: Readiness trends - sleep regularity | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of physical readiness trends, including sleep regularity - a measure of consistency of bedtime, wake-time and duration sleep over a period of time.
Oura Ring Sleep Data: Readiness trends - readiness score | Oura data is collected from daily wear of ring from date of randomization through study completion after 3 weeks.
  Oura Ring will continuously measure aspects of physical readiness trends, including readiness score - calculated from multiple other aspects of sleep data and readiness trends.

OTHER OUTCOMES:
Body Measurements: Height (cm) | Measured prior to treatment starting at time of enrollment.
  Biometrics
Body Measurements: Weight (kg/lbs) | Measured prior to treatment starting at time of enrollment.
  Biometrics
Body Measurements: Body composition (% body fat) | Measured prior to treatment starting at time of enrollment.
  Biometrics
Body Measurements: C1 - proximal thigh circumference (cm) | Measured prior to treatment starting at time of enrollment.
  Biometrics - used to calculate PBMT dosage
Body Measurements: C2 - distal thigh circumference (cm) | Measured prior to treatment starting at time of enrollment.
  Biometrics - used to calculate PBMT dosage
Body Measurements: L1 - length of thigh (cm) | Measured prior to treatment starting at time of enrollment.
  Biometrics - used to calculate PBMT dosage

CONTACTS AND LOCATIONS:
Overall Officials: Bradley H Cornell, DPT, Principal Investigator — 1st Special Forces Group Tactical Human Optimization, Rapid Rehabilitation and Reconditioning (THOR3)
Locations (1):
- Joint Base Lewis-McChord, Joint Base Lewis McChord, Washington, United States

IPD SHARING:
Plan to Share IPD: Yes
The Initial Consent Form (ICF) for this research study states that de-identified research data will be shared with MIRROR and USU and maintained indefinitely for possible use in future research. By consenting to participate in this research study, participants agree to allow us to maintain their de-identified research data indefinitely for possible use in future research.
  Participants will not be given the option to opt out of us retaining their de-identified research data indefinitely for possible future use. The ICF states, "If you do not want your deidentified data collected as part of this research study to be kept for use in future research studies, you should not sign this consent form."
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Ailioaie LM, Litscher G. Photobiomodulation and Sports: Results of a Narrative Review. Life (Basel). 2021 Dec 3;11(12):1339. doi: 10.3390/life11121339. PMID 34947870
- [Background] Antonialli FC, De Marchi T, Tomazoni SS, Vanin AA, dos Santos Grandinetti V, de Paiva PR, Pinto HD, Miranda EF, de Tarso Camillo de Carvalho P, Leal-Junior EC. Phototherapy in skeletal muscle performance and recovery after exercise: effect of combination of super-pulsed laser and light-emitting diodes. Lasers Med Sci. 2014 Nov;29(6):1967-76. doi: 10.1007/s10103-014-1611-7. Epub 2014 Jun 19. PMID 24942380
- [Background] Aver Vanin A, De Marchi T, Tomazoni SS, Tairova O, Leao Casalechi H, de Tarso Camillo de Carvalho P, Bjordal JM, Leal-Junior EC. Pre-Exercise Infrared Low-Level Laser Therapy (810 nm) in Skeletal Muscle Performance and Postexercise Recovery in Humans, What Is the Optimal Dose? A Randomized, Double-Blind, Placebo-Controlled Clinical Trial. Photomed Laser Surg. 2016 Oct;34(10):473-482. doi: 10.1089/pho.2015.3992. Epub 2016 Aug 29. PMID 27575834
- [Background] Baroni BM, Leal Junior EC, De Marchi T, Lopes AL, Salvador M, Vaz MA. Low level laser therapy before eccentric exercise reduces muscle damage markers in humans. Eur J Appl Physiol. 2010 Nov;110(4):789-96. doi: 10.1007/s00421-010-1562-z. Epub 2010 Jul 3. PMID 20602109
- [Background] Baroni BM, Rodrigues R, Freire BB, Franke Rde A, Geremia JM, Vaz MA. Effect of low-level laser therapy on muscle adaptation to knee extensor eccentric training. Eur J Appl Physiol. 2015 Mar;115(3):639-47. doi: 10.1007/s00421-014-3055-y. Epub 2014 Nov 23. PMID 25417170
- [Background] Vieira WH, Ferraresi C, Perez SE, Baldissera V, Parizotto NA. Effects of low-level laser therapy (808 nm) on isokinetic muscle performance of young women submitted to endurance training: a randomized controlled clinical trial. Lasers Med Sci. 2012 Mar;27(2):497-504. doi: 10.1007/s10103-011-0984-0. Epub 2011 Aug 26. PMID 21870127
- [Background] de Carvalho G, Gobbi A, Gobbi RB, Alfredo DMN, do Carmo Furquim TH, Barbosa RI, Papoti M, de Jesus Guirro RR. Photobiomodulation by light emitting diode applied sequentially does not alter performance in cycling athletes. Lasers Med Sci. 2020 Oct;35(8):1769-1779. doi: 10.1007/s10103-020-02973-9. Epub 2020 Feb 20. PMID 32078062
- [Background] De Marchi T, Leal-Junior ECP, Lando KC, Cimadon F, Vanin AA, da Rosa DP, Salvador M. Photobiomodulation therapy before futsal matches improves the staying time of athletes in the court and accelerates post-exercise recovery. Lasers Med Sci. 2019 Feb;34(1):139-148. doi: 10.1007/s10103-018-2643-1. Epub 2018 Sep 27. PMID 30264178
- [Background] de Oliveira AR, Vanin AA, Tomazoni SS, Miranda EF, Albuquerque-Pontes GM, De Marchi T, Dos Santos Grandinetti V, de Paiva PRV, Imperatori TBG, de Carvalho PTC, Bjordal JM, Leal-Junior ECP. Pre-Exercise Infrared Photobiomodulation Therapy (810 nm) in Skeletal Muscle Performance and Postexercise Recovery in Humans: What Is the Optimal Power Output? Photomed Laser Surg. 2017 Nov;35(11):595-603. doi: 10.1089/pho.2017.4343. PMID 29099680
- [Background] de Paiva PR, Tomazoni SS, Johnson DS, Vanin AA, Albuquerque-Pontes GM, Machado CD, Casalechi HL, de Carvalho PT, Leal-Junior EC. Photobiomodulation therapy (PBMT) and/or cryotherapy in skeletal muscle restitution, what is better? A randomized, double-blinded, placebo-controlled clinical trial. Lasers Med Sci. 2016 Dec;31(9):1925-1933. doi: 10.1007/s10103-016-2071-z. Epub 2016 Sep 13. PMID 27624781
- [Background] Dompe C, Moncrieff L, Matys J, Grzech-Lesniak K, Kocherova I, Bryja A, Bruska M, Dominiak M, Mozdziak P, Skiba THI, Shibli JA, Angelova Volponi A, Kempisty B, Dyszkiewicz-Konwinska M. Photobiomodulation-Underlying Mechanism and Clinical Applications. J Clin Med. 2020 Jun 3;9(6):1724. doi: 10.3390/jcm9061724. PMID 32503238
- [Background] Dornelles MP, Fritsch CG, Sonda FC, Johnson DS, Leal-Junior ECP, Vaz MA, Baroni BM. Photobiomodulation therapy as a tool to prevent hamstring strain injuries by reducing soccer-induced fatigue on hamstring muscles. Lasers Med Sci. 2019 Aug;34(6):1177-1184. doi: 10.1007/s10103-018-02709-w. Epub 2019 Jan 3. PMID 30607719
- [Background] Faul F, Erdfelder E, Lang AG, Buchner A. G*Power 3: a flexible statistical power analysis program for the social, behavioral, and biomedical sciences. Behav Res Methods. 2007 May;39(2):175-91. doi: 10.3758/bf03193146. PMID 17695343
- [Background] Ferraresi C, Dos Santos RV, Marques G, Zangrande M, Leonaldo R, Hamblin MR, Bagnato VS, Parizotto NA. Light-emitting diode therapy (LEDT) before matches prevents increase in creatine kinase with a light dose response in volleyball players. Lasers Med Sci. 2015 May;30(4):1281-7. doi: 10.1007/s10103-015-1728-3. Epub 2015 Feb 27. PMID 25722067
- [Background] Ferraresi C, Bertucci D, Schiavinato J, Reiff R, Araujo A, Panepucci R, Matheucci E Jr, Cunha AF, Arakelian VM, Hamblin MR, Parizotto N, Bagnato V. Effects of Light-Emitting Diode Therapy on Muscle Hypertrophy, Gene Expression, Performance, Damage, and Delayed-Onset Muscle Soreness: Case-control Study with a Pair of Identical Twins. Am J Phys Med Rehabil. 2016 Oct;95(10):746-57. doi: 10.1097/PHM.0000000000000490. PMID 27088469
- [Background] Hamblin MR. Shining light on the head: Photobiomodulation for brain disorders. BBA Clin. 2016 Oct 1;6:113-124. doi: 10.1016/j.bbacli.2016.09.002. eCollection 2016 Dec. PMID 27752476
- [Background] Leal Junior EC, de Godoi V, Mancalossi JL, Rossi RP, De Marchi T, Parente M, Grosselli D, Generosi RA, Basso M, Frigo L, Tomazoni SS, Bjordal JM, Lopes-Martins RA. Comparison between cold water immersion therapy (CWIT) and light emitting diode therapy (LEDT) in short-term skeletal muscle recovery after high-intensity exercise in athletes--preliminary results. Lasers Med Sci. 2011 Jul;26(4):493-501. doi: 10.1007/s10103-010-0866-x. Epub 2010 Nov 19. PMID 21088862
- [Background] Leal Junior EC, Lopes-Martins RA, Baroni BM, De Marchi T, Rossi RP, Grosselli D, Generosi RA, de Godoi V, Basso M, Mancalossi JL, Bjordal JM. Comparison between single-diode low-level laser therapy (LLLT) and LED multi-diode (cluster) therapy (LEDT) applications before high-intensity exercise. Photomed Laser Surg. 2009 Aug;27(4):617-23. doi: 10.1089/pho.2008.2350. PMID 19302015
- [Background] Pinto HD, Vanin AA, Miranda EF, Tomazoni SS, Johnson DS, Albuquerque-Pontes GM, Aleixo IO Junior, Grandinetti VD, Casalechi HL, de Carvalho PT, Leal-Junior EC. Photobiomodulation Therapy Improves Performance and Accelerates Recovery of High-Level Rugby Players in Field Test: A Randomized, Crossover, Double-Blind, Placebo-Controlled Clinical Study. J Strength Cond Res. 2016 Dec;30(12):3329-3338. doi: 10.1519/JSC.0000000000001439. PMID 27050245
- [Background] Rossato M, Dellagrana RA, Sakugawa RL, Baroni BM, Diefenthaeler F. Dose-Response Effect of Photobiomodulation Therapy on Muscle Performance and Fatigue During a Multiple-Set Knee Extension Exercise: A Randomized, Crossover, Double-Blind Placebo-Controlled Trial. Photobiomodul Photomed Laser Surg. 2020 Dec;38(12):758-765. doi: 10.1089/photob.2020.4820. Epub 2020 Nov 24. PMID 33232629
- [Background] Tomazoni SS, Machado CDSM, De Marchi T, Casalechi HL, Bjordal JM, de Carvalho PTC, Leal-Junior ECP. Infrared Low-Level Laser Therapy (Photobiomodulation Therapy) before Intense Progressive Running Test of High-Level Soccer Players: Effects on Functional, Muscle Damage, Inflammatory, and Oxidative Stress Markers-A Randomized Controlled Trial. Oxid Med Cell Longev. 2019 Nov 16;2019:6239058. doi: 10.1155/2019/6239058. eCollection 2019. PMID 31827687
- [Background] Vanin AA, Miranda EF, Machado CS, de Paiva PR, Albuquerque-Pontes GM, Casalechi HL, de Tarso Camillo de Carvalho P, Leal-Junior EC. What is the best moment to apply phototherapy when associated to a strength training program? A randomized, double-blinded, placebo-controlled trial : Phototherapy in association to strength training. Lasers Med Sci. 2016 Nov;31(8):1555-1564. doi: 10.1007/s10103-016-2015-7. Epub 2016 Jul 1. PMID 27371449
- [Background] Wyatt Daniel Army Staff SGT. Program boosts special forces members' physical, mental capabilities. U.S. Department of Defense. December 6, 2017. Accessed July 13, 2022. https://www.defense.gov/News/News-Stories/Article/Article/1389545/program-boosts-specialforces- members-physical-mental-capabilities/
- See also: Homepage for all current Photomedicine projects, including PM#14. — https://mirrorusuhs.org/photomedicine-research

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2024-03-20): https://cdn.clinicaltrials.gov/large-docs/79/NCT06380179/Prot_SAP_000.pdf
  • Informed Consent Form (2024-03-19): https://cdn.clinicaltrials.gov/large-docs/79/NCT06380179/ICF_001.pdf